CLINICAL TRIAL: NCT07253662
Title: Phase I Trial of Pressurized Intraperitoneal Aerosolized Chemotherapy (PIPAC) in Patients With Peritoneal Metastasis From Pancreatic Adenocarcinoma
Brief Title: Pressurized Intraperitoneal Aerosolized Chemotherapy (PIPAC) in Patients With Peritoneal Metastasis From Pancreatic Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0087
Record Dates: First submitted 2025-09-26; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Adenocarcinoma Pancreas
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): This study is a prospective single center, non-randomized phase I trial to confirm the safety of PIPAC with nab- paclitaxel in conjunction with standard of care systemic therapy in patients with peritoneal-only metastasis from PDAC. The efficacy signals noted in this trial will inform a potential phase II/III multicenter clinical trial.
  Patients may receive up to 3 treatments whilst enrolled on the study, with a potential opportunity to extend outside of the trial for compassionate use.
  Interventions: Device: PIPAC; Drug: Nab-paclitaxel

INTERVENTIONS:
Device: PIPAC — Pressurized Intra Peritoneal Aerosol Chemotherapy (PIPAC) is a novel therapeutic approach that is minimally invasive, does not require cytoreduction (laparotomy) and can be frequently repeated. PIPAC entails accessing the abdominal cavity using standard laparoscopic techniques with the chemotherapeutics aerosolized via a high-pressure micro-injection pump (MIP) . PIPAC has not yet been investigated in the US and remains investigational in Europe. A MIP is utilized to aerosolize and deliver chemotherapeutic medications into the abdominal cavity during laparoscopy for treatment of primary and secondary peritoneal malignancy. The study device consists of a nebulizer, that when connected to a high-pressure injector, is inserted into the abdomen during a laparoscopic procedure. Pressurization of the liquid chemotherapy through the study device results in aerosolization of the chemotherapy intra-abdominally. The device is single use and not re-sterilized. It is removed at the conclusion
Drug: Nab-paclitaxel — The dose for this intervention will be 112.5mg/m2, for which the rationale is provided in section 4.3: Justification of Dose. Nab-paclitaxel will be delivered during the PIPAC procedures via the device described above over 5 minutes and will remain in contact with the peritoneum for 30 minutes, after which the pneumoperitoneum will be evacuated, and the abdomen closed. Nab-paclitaxel is diluted in total volume of 200 ml NaCl 0.9%. The solution will be used within 4 hours of reconstitution per prescribing recommendation (if longer, a new solution will be reconstituted). This will be repeated twice, every six weeks, for a total of three PIPAC procedures.

SUMMARY:
Palliative systemic therapy is the standard treatment option for patients with pancreatic ductal adenocarcinoma (PDAC) and peritoneal metastasis (PM), who have a median overall survival of only 6-11 months and a serious adverse event (SAE) rate of >5%. Patients with peritoneal-only metastasis may demonstrate unique tumor biology with less potential for hematogenous and lymphatic spread, making them potential candidates for a regional approach directed at the peritoneum. PIPAC is a drug- delivery system that combines the pharmacokinetic advantages of low- dose intraperitoneal chemotherapy (high tumor tissue penetration with low systemic absorption/toxicity) with the principles of aerosolization (homogenous intraperitoneal distribution and deeper tissue penetration). PIPAC may offer a complimentary approach to maximize drug delivery to tumor implants, potentially improving quality of life and survival without significant additional morbidity. Several non-randomized studies have evaluated safety, feasibility, and efficacy of PIPAC with various intraperitoneal agents in a variety of tumor types. Very few patients with pancreatic cancer PM have been included in these studies and most have been treated with either PIPAC-oxaliplatin or doxorubicin/cisplatin. A recent phase 1 dose-escalation study included patients with ovarian, gastric, breast, and hepatopancreatobiliary malignancies. One patient with

pancreatic cancer was included in this study. The recommended phase 2 dose was 140 mg/m2, with guidance to decrease the dose to 112.5 mg/m2 in patients with hepatic impairment. Therefore, the dose utilized in this study is 112.5 mg/m2. This recommendation was based on concern for nab-paclitaxel hepatotoxicity, but there was no data presented to support this expert recommendation.

This study sets out to explore the role of PIPAC with nab-paclitaxel in combination with medical oncology choice standard of care therapy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign informed consent form
* Age ≥18 years
* Patient must have histologically confirmed pancreatic adenocarcinoma with either histologic confirmation or strong suspicion of peritoneal metastasis on cross sectional imaging
* ECOG performance status ≤ 2
* Pre-treatment Laboratory Parameters:
* Absolute neutrophil count (ANC) > 1500/mm3
* Platelets > 100,000/mm3
* Hemoglobin > 9 g/dl
* Serum total bilirubin < 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN, unless patient is known to have chronic liver disease (hepatitis) in which case AST and ALT must be ≤ 5 x ULN.
* Creatinine clearance (Ccr) > 40 ml/min

  * No contraindications for a laparoscopy.
* The peritoneal disease does not have to be measurable by RECIST 1.1 but needs to visible on cross sectional imaging or diagnostic laparoscopy.
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Women of childbearing potential (WOCBP) and male patients with WOCBP partner must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 6 months after the PIPAC or last dose of chemotherapy in such a manner that the risk of pregnancy is minimized .-WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post menopause is defined as:

Amenorrhea ≥ 12 consecutive months without another cause or For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered of childbearing potential.

Inclusion to proceed with PIPAC :

Laparoscopy findings must meet all of the below criteria in order to proceed to PIPAC:

* PIPAC access is feasible
* There is room for aerosol therapy
* There is no evidence of impending bowel obstruction
* < 5 L of ascites
* Not a candidate for cytoreduction and HIPEC

Exclusion Criteria:

* Confirmed or suspected extra-peritoneal metastasis
* Bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy or exclusive total parenteral nutrition.
* Life expectancy of less than 4 months.
* Prior intra-abdominal aerosol chemotherapy
* Previous anaphylactic reaction to the nab-paclitaxel drug used.
* Intra-abdominal Ascites >5L
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias, severe renal impairment, myelosuppression, or severe hepatic impairment.
* Immunocompromised patients such as those with an immunosuppressive medication or a known disease of the immune system.
* New York Heart Association (NYHA) Class 3 or 4; myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months.
* Exclusive total parenteral nutrition.
* Pregnancy. Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
To confirm the safety and tolerability of PIPAC with nab-paclitaxel in conjunction with medical oncologist choice standard of care therapy with CTCAE v5.0 | 2 years
  DLTs are defined as any of the following events (based on CTCAE v5 and Clavien Dindo) during the first PIPAC cycle and attributable to PIPAC:
  Any grade 3 or 4 non-hematologic toxicity, excluding:
  Grade 3 nausea, vomiting, abdominal pain, or diarrhea that is adequately treated to grade 2 or lower within 48 hours.
  Grade 3 fatigue that returns to grade 2 or less within 7 days.
  Grade 3 laboratory/metabolic abnormalities that are not considered clinically significant or are easily correctable to grade 2 or lower within 72 hours.
  Grade 3 infusion-related reaction (first occurrence and in the absence of steroid prophylaxis) that resolves within 6 hours with appropriate clinical management.
  Grade 3 peripheral neuropathy
  Surgical complication of Clavien-Dindo grade IIIB or greater
To confirm the safety and tolerability of PIPAC with nab-paclitaxel in conjunction with medical oncologist choice standard of care therapy. Measurement of AEs according to NCI CTCAE version 5.0 during the first cycle, or throughout the 6 weeks following | 2 years
  Safety: DLTs during the safety evaluation period (6 weeks after initial PIPAC)
  DLTs are defined as any of the following events (based of CTCAE v5 and Clavien Dindo) during the first PIPAC cycle and attributable to PIPAC:
  Any Grade 3 laboratory/metabolic abnormality that requires medical intervention, irrespective of the duration of the event
  Any grade 3 or 4 non-hematologic toxicity excluding:
  Grade 3 treated nausea, vomiting, abdominal pain, or diarrhea that is adequately treated to grade 2 or lower within 48 hours.
  Grade 3 fatigue that returns to grade 2 or less within 7 days.
  Grade 3 laboratory/metabolic abnormalities that are not considered clinically significant or are easily correctable to grade 2 or lower within 72 hours.
  Grade 3 infusion related reaction (first occurrence and in the absence of steroid prophylaxis) that resolves within 6 hours with appropriate clinical management.
  Grade 3 peripheral neuropathy
  Surgical complication of Clavien-Dindo grade IIIB

OTHER OUTCOMES:
Safety/tolerability | 2 years
  To assess the efficacy/anti-tumoral activity, feasibility/ compliance, further assessment of safety and tolerability, as well as overall and progression-free survival, quality of life, and pharmacokinetics of PIPAC-nab-paclitaxel on disease progression Number of patients with severe (greater than or equal to grade 3 CTC AEs throughout the study [beyond the 6-week DLT period for PIPAC 1]) including any long-term toxicity attributable to PIPAC
  Number of patients with minor toxicity, defined as CTCAE grade 2 or less during the treatment period
Post-operative surgical complications by Clavien-Dindo during the trial period. | 2 years
  This will be measured using the Clavien Dindo scale
Efficacy/ Anti-tumoral Response | 2 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228- 247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside the Northwell institution.